CLINICAL TRIAL: NCT04922099
Title: Glycemic Gap Versus Admission Plasma Glucose Level As Predictors of ICU Out Comes in Type 2 Diabetic Patients With Acute Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatema Medhat Ahmed, resident doctor, Assiut University
Other Study IDs: Glycemic gap
Record Dates: First submitted 2021-05-25; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Assess the Relation Between Glycemic Gab and Adverse Clinical Outcomes in Diabetic Patients Who Hospitalized With Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: glycemic gap — Measurements of HbA1c-based adjusted glycemic gap:
  The estimated chronic average glucose levels (eAG) over the past 3 months will calculate from the equation AG = 28.7 × HbA1c - 46.7 Glycemic gap was calculated as the ADAG level subtracted from the admission glucose level.

SUMMARY:
assess the relation between glycemic gab and adverse clinical outcomes in diabetic patients who hospitalized with heart failure

DETAILED DESCRIPTION:
Hyperglycemia is a common problem in patients wi9non-diabetic patients but not in patients with diabetes . The relationship between admission hyperglycemia and mortality in diabetic patients with AHF or critical illness remains controversial . Those discrepancies could be partly attributed to long-term glycemic control in diabetic patients.

Critical illness can induce stress-induced hyperglycemia (SIH), which results from the excess release of counter-regulatory hormones and anti-inflammatory cytokines, leading to augmented gluconeogenesis and insulin resistance.

In diabetic patients with acute illness, the phenomenon of admission hyperglycemia could be connected with acute physiological stress, poorer glycemic controls, or a combination of both . It is necessary to think about background glycemic control when exploring the relationships between admissions Hyperglycemia and clinical outcomes. Recent studies have shown that hemoglobin A1c (HbA1c)-based adjusted glycemic variables, including glycemic gap and stress hyperglycemia ratio, were linked to severity of disease and unfavorable prognosis in diabetic patients with some infectious diseases, cardiovascular diseases and clinical illness

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients admitted to ICU of internal medicine department from October 2020 to November 2021 by heart failure

Exclusion Criteria:

* Age ≤18 years.

  1. Hypoglycemia (plasma glucose <70 mg/dL) at initial presentation.
  2. An admission diagnosis of diabetic ketoacidosis or hyperosmolar hyperglycemic state.
  3. Patients with hemoglobin variants (e.g., sickle cell anemia, thalassemia) or with hematologic conditions (e.g., hemolytic anemia) that could interfere with the accuracy of the HbA1c assay.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All diabetic patients admitted to ICU of internal medicine department from October 2020 to November 2021 by heart failure
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic gap versus admission plasma glucose level As predictors of ICU out comes in type 2 diabetic patients with acute heart failure | through study completion an avarage 1 year
  Glycemic gap versus admission plasma glucose level As predictors of ICU out comes in type 2 diabetic patients with acute heart failure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lazzeri C, Valente S, Chiostri M, D'Alfonso MG, Spini V, Angelotti P, Gensini GF. Admission Glycaemia and Acute Insulin Resistance in Heart Failure Complicating Acute Coronary Syndrome. Heart Lung Circ. 2015 Nov;24(11):1074-80. doi: 10.1016/j.hlc.2015.04.171. Epub 2015 May 16. PMID 26031570
- [Background] de Miguel-Yanes JM, Gonzalo-Hernando C, Munoz-Rivas N, Mendez-Bailon M, Cava-Valenciano F, Torres-Macho J. First plasma glucose value after urgent admission and in-hospital mortality in acutely decompensated heart failure. Heart Lung. 2015 Mar-Apr;44(2):137-40. doi: 10.1016/j.hrtlng.2014.11.006. Epub 2014 Dec 18. PMID 25534479
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235
- [Background] Yang CJ, Liao WI, Wang JC, Tsai CL, Lee JT, Peng GS, Lee CH, Hsu CW, Tsai SH. Usefulness of glycated hemoglobin A1c-based adjusted glycemic variables in diabetic patients presenting with acute ischemic stroke. Am J Emerg Med. 2017 Sep;35(9):1240-1246. doi: 10.1016/j.ajem.2017.03.049. Epub 2017 Mar 22. PMID 28363620